CLINICAL TRIAL: NCT05689086
Title: A Virtual Heart Failure Optimization Program for Guideline Directed Medical Therapy and Cardiac Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge Cardiac Care Centre (Other)
Responsible Party: Sponsor
Other Study IDs: CCCiCHF20
Record Dates: First submitted 2022-12-13; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Program Participants: Patients with HFrEF (LVEF<40%) & NYHA class II-III who are referred to and consent to participate in the "Virtual Heart Failure Optimization Program"
  Interventions: Other: Virtual Heart Failure Optimization Program

INTERVENTIONS:
Other: Virtual Heart Failure Optimization Program — Participants referred to the "Virtual Heart Failure Optimization Program" will be seen for initial consultation by a HF program nurse and cardiologist within 1 week. Patients will be offered the opportunity to participate in virtual cardiac rehabilitation.
  Following this, patients will be assessed virtually every two weeks by a HF program nurse for addition and up-titration of medical therapy. All medication changes will be performed algorithmically and reviewed with the overseeing cardiologist. Following all medication changes, appropriate monitoring will be performed algorithmically as well.
  All participants will be asked if they would like to participate in cardiac rehabilitation and an automatic referral will be sent by the overseeing cardiologist. Virtual cardiac rehabilitation will be conducted weekly with phone follow-up appointments with a program kinesiologist and virtual education programming.

SUMMARY:
The goal of this study is to test the impact of a virtual heart failure optimization program on uptake of guideline directed medical therapy, participation in cardiac rehabilitation & impact on echocardiographic parameters.

DETAILED DESCRIPTION:
This is a single center, prospective pre-post cohort study testing a virtual, multi-disciplinary heart failure optimization program for up-titration of guideline directed medical therapy. This nurse and kinesiologist-led program will start and up-titrate patients on GDMT and offer virtual cardiac rehabilitation over a 3-month period.

The investigators hypothesize that this program could safely achieve higher rates of maximally tolerated ARNI, Beta-blocker, MRA and SGLT2i rates, as well as participation in cardiac rehabilitation among HFrEF patient participants. The investigators hypothesize that participation will lead to improved Left Ventricular Ejection Fraction on Echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* HFrEF (ejection fraction less than 40%) with New York Heart Association (NYHA) class II or III symptoms
* Adults (>18 years of age), capable of providing informed consent, English-proficient and with access to a telephone

Exclusion Criteria:

* Patients who are pregnant
* Patients who who are incarcerated
* Cardiac Transplant Patients
* Patients with Left Ventricular Assist Devices

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with HFrEF (ejection fraction less than 40%) with New York Heart Association (NYHA) class II or III symptoms
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Doses of GDMT | After completion of program (3 months)
  Beta-blocker, ACE-inhibitor/Angiotensin receptor blocker/Valsartan-Sacubitril, Mineralocorticoid Receptor Antagonist, SGLT2 inhibitor
Change from baseline Left Ventricular Ejection Fraction | After completion of program (3 months)
  Measured in Transthoracic Echocardiogram

SECONDARY OUTCOMES:
Change from baseline NYHA Classification | After completion of program (3 months)
  Stage of Heart Failure (I-IV, IV is worse)
Change from baseline Left Ventricular Mass Index | After completion of program (3 months)
  Measured by Transthoracic Echocardiogram
Change from baseline Left Ventricular End Diastolic Diameter | After completion of program (3 months)
  Measured by Transthoracic Echocardiogram
Change from baseline Left Ventricular End Systolic Diameter | After completion of program (3 months)
  Measured by Transthoracic Echocardiogram
Change from baseline Serum Potassium | After completion of program (3 months)
Change from baseline eGFR | After completion of program (3 months)
Change from baseline Systolic Blood Pressure | After completion of program (3 months)
Change from baseline Diastolic Blood Pressure | After completion of program (3 months)
Change from baseline Heart Rate | After completion of program (3 months)
Change from baseline Body Mass Index | After completion of program (3 months)

CONTACTS AND LOCATIONS:
Overall Officials: A. Pandey, MD, Study Chair — Cambridge Cardiac Care Centre
Locations (1):
- Cambridge Cardiac Rehab, Cambridge, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No